CLINICAL TRIAL: NCT05640999
Title: A Phase II Study of Tailored Adjuvant Therapy in POLE-Mutated and p53-Wildtype/NSMP Early Stage Endormetrial Cancer (RAINBO BLUE & TAPER)
Brief Title: Adjuvant Therapy in POLE-Mutated and p53-Wildtype/NSMP Early Stage Endometrial Cancer RAINBO BLUE & TAPER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Cancer Clinical Trials Network (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN10; NRG-GY032 (Other: NRG); NCT06388018 (obsolete NCT alias)
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiotherapy, Adjuvant; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Sub-study A: RAINBO BLUE Cohort A1 (Experimental): Observation
  Interventions: Other: Observation
- Sub-Study A: RAINBO BLUE Cohort A2 (Experimental): Observation or Adjuvant Radiotherapy
  Interventions: Radiation: Adjuvant radiotherapy (EBRT +/- brachytherapy); Other: Observation
- Sub-Study B: TAPER (Experimental): Observation or Vaginal Brachytherapy
  Interventions: Radiation: Vaginal brachytherapy; Other: Observation

INTERVENTIONS:
Radiation: Vaginal brachytherapy — Vaginal brachytherapy should be delivered using a vaginal cylinder, or alternatively ovoids
  Arms: Sub-Study B: TAPER
Radiation: Adjuvant radiotherapy (EBRT +/- brachytherapy) — Treatment is to be delivered using 4-18 MV photons. MV, kV or CBCT imaging capabilities are required. Planning systems with capability for DICOM data transfer must be used.
  Arms: Sub-Study A: RAINBO BLUE Cohort A2
Other: Observation — Observation

SUMMARY:
This protocol tests de-escalated adjuvant treatment in patients with POLE-mutated or p53wt/NSMP (p53 wildtype/no specific molecular profile) early-stage endometrial cancer (EC). Patients may be enrolled in one of two sub-studies

* EN10.A/RAINBO BLUE: POLE-mutated EC
* EN10.B/TAPER: p53 wildtype / NSMP EC

DETAILED DESCRIPTION:
This study is being done in order to find out if this new approach is better or worse than the usual approach for early-stage endometrial cancer. The usual approach is defined as the care most people get for early-stage endometrial cancer.

The usual approach for patients who are not in a study is treatment with surgery. Tissue that is removed as part of this procedure is analyzed in the pathology laboratory to guide the doctor to decide whether or not additional treatment such as radiation and or chemotherapy should be recommended.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had surgery consisting of hysterectomy and bilateral salpingo-oophorectomy. Lymph node dissection can be performed as per institutional standards. There must be no macroscopic residual disease after surgery.
* Patients must have histologically confirmed Stage I to III endometrial carcinoma which can be endometrioid, serous, clear cell, un/dedifferentiated, carcinosarcoma or mixed.
* Patients' Eastern Cooperative Group (ECOG) performance status must be 0, 1, or 2.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients' age must be ≥ 18 years.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Patient is able (i.e. sufficiently fluent) and willing to complete the patient-reported outcomes (PRO) questionnaires in either English, French or a validated language
* Patients must be accessible for treatment and follow-up. Patients enrolled on this trial must be treated and followed at the participating centre
* Protocol treatment is to begin within 10 weeks of hysterectomy/bilateral salpingo-oophorectomy

Exclusion Criteria:

* Prior Neoadjuvant chemotherapy for current endometrial cancer diagnosis.
* Prior pelvic radiation.
* Patients with a history of other malignancies, except: carcinoma in-situ without evidence of invasive disease when resected, adequately treated non-melanoma skin cancer, or other tumours curatively treated with no evidence of disease for ≥ 5 years.
* Clinical evidence of distant metastasis as determined by pre-surgical or post-surgical imaging (CT scan of chest, abdomen and pelvis or whole-body PET-CT scan)
* Patients with a documented positive surgical margin.
* Patients with a documented positive peritoneal washings, if performed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 393 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Estimate the rate of pelvic recurrence at 3 years in patients who are treated with de-escalated adjuvant treatment directed by tumour molecular status | 3 years

SECONDARY OUTCOMES:
Estimate the rate of isolated vaginal recurrence at 3 years | 3 years
Estimate the rate of para-aortic recurrence at 3 years | 3 years
Estimate the rate of distant metastasis at 3 years | 3 years
Estimate recurrence-free survival | 9 years
Estimate endometrial cancer-specific survival | 9 years
Estimate overall survival | 9 years
Describe the impact of molecular classification on fear of recurrence by Fear of Recurrence Inventory | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Han, Study Chair — University Health Network, Princess Margaret Hospital, Toronto ON Canada; Jessica McAlpine, Study Chair — BCCA-Vancouver Cancer Centre, Vancouver BC Canada
Locations (96):
- United States (60):
  - Alaska Womens Cancer Care, Anchorage, Alaska
  - University of Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Huntington Memorial Hospital, Pasadena, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Sarasota Memorial Hospital - Venice, N. Venice, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - First Physicians Group-Sarasota, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Sarasota Memorial Health Care Centre, Sarasota, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Josephs Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Centre, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Womens Cancer Center of Nevada, Las Vegas, Nevada
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Upstate Cancer Center Radiation Oncology at Oswego, Oswego, New York
  - State University of New York, Syracuse, New York
  - Upstate Cancer Center at Hill Radiation Oncology, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Womens Cancer Care Raleigh, Raleigh, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Centre, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - M.D. Anderson Cancer Center, Houston, Texas
  - Farmington Health Centre, Farmington, Utah
  - University of Utah Sugarhouse Health Centre, Salt Lake City, Utah
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center First Hill, Seattle, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - South Western Sydney Local Health District, Liverpool, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Research Institute South Brisbane, South Brisbane, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Frankston Hospital, Frankston, Victoria
  - The Royal Women's Hospital, Parkville, Victoria
  - Canberra Hospital, Garran
  - Royal Brisbane and Womens Hospital, Herston
- Canada (14):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA - Prince George, Prince George, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - BCCA - Victoria, Victoria, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec
- France (3):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Institut Gustave-Roussy, Villejuif, FR
  - Institut Universitaire du Cancer de Toulouse - IUCT, Toulouse, Occitanie
- Italy (2):
  - ASST Spedali Civili Brescia, Brescia
  - European Institute of Oncology, Milan
- Netherlands (6):
  - Radiotherapiegroep, Arnhem, Gelderland
  - Maastro clinic (Maastricht UMC), Maastricht, Limburg
  - Catharina ziekenhuis, Eindhoven, North Brabant
  - MC Haaglanden, The Hague, South Holland
  - Erasmus Medical Center (EMC), Rotterdam, The Netherlands
  - Leiden University Medical Center (LUMC), Leiden
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: No